CLINICAL TRIAL: NCT05493748
Title: Virtual Bladder Training for Overactive Bladder Syndrome in Women. Which Symptom Responds Better?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, AGUSTINA VENDRAMINI, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: # 6237 PRIISA 6017
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder Syndrome; Bladder Training

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, before-after trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frequency (Other): Main symptom: Increased daytime urinary frequency: complaint that micturition occurs more frequently during waking hours than previously deemed normal by the woman.
  Interventions: Other: Bladder training
- Nocturia (Other): Main symptom: Complaint of interruption of sleep one or more times because of the need to micturate.
  Interventions: Other: Bladder training

INTERVENTIONS:
Other: Bladder training — Bladder training for overactive bladder syndrome.

SUMMARY:
According to International Urogynecological Association and International Continence Society joint report on the terminology for female pelvic floor dysfunction, overactive bladder syndrome (OAB) is defined as urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of urinary tract infection or other obvious pathology. Bladder training lasting for a minimum of 4 to 6 weeks is indicated as a first-line treatment. The investigators' goal is to compare changes in satisfaction, measured in terms of quality of life, in 2 groups of women with different main accompanying symptoms in OAB (frequency vs. nocturia), before and after bladder training utilizing telemedicine (virtual bladder training), for 4 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years of age
* Live in Buenos Aires City
* Overactive Bladder Syndrome
* Access to virtual appointment

Exclusion Criteria:

* Previous overactive bladder syndrome treatment.
* Prior stress urinary incontinence or pelvic organ prolapse surgery.
* History of Neurogenic Bladder, pelvic organs prolapse or pelvic radiation.
* Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in King's Health Questionnaire (KHQ) score | Change from Baseline King's Health Questionnaire at 6 weeks
  KHQ score: 0-100 points per domain. Higher scores mean a worse outcome.Ten points change in KHQ score, before and after bladder training.
Change in International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) score | Change from Baseline International Consultation on Incontinence Questionnaire Short Form at 6 weeks
  ICIQ SF score: 0-21 points. Higher scores mean a worse outcome. Three points change in ICIQ-SF score, before and after bladder training.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina